CLINICAL TRIAL: NCT04514692
Title: Phase 1-2 Study of Individualized Bone Marrow Sparing Image Guided Radiotherapy Incorporating Novel Use of Granulocyte Colony Stimulating Factor and FDG PET Imaging
Brief Title: Bone Marrow Sparing Image-Guided Radiation Therapy (RT) Incorporating Novel Use of GCSF and FDG-PET Imaging
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Elizabeth Kidd, Associate Professor of Radiation Oncology (Radiation Therapy), Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-56842; GYN0007 (Other: OnCore); NCI-2021-03444 (Registry Identifier: NCI- Clinical Trials Reporting Program)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-02

CONDITIONS: Cervix Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase I -Dose finding, Cohort 1 (Experimental): Dosing will occur in cohorts of 3 patients with the start at dose of GCSF will be 780 mcg x 3 days
  Interventions: Drug: GCSF
- Phase I -Dose finding, Cohort 2 (Experimental): Dosing will occur in cohorts of 3 patients, If 3 out of 3 patients achieve the target SUVmean, the GCSF dose will be 780 mcg x 2 days
  Interventions: Drug: GCSF
- Phase I -Dose finding, Cohort 3 (Experimental): Dosing will occur in cohorts of 3 patients, If 3 out of 3 patients achieve the target SUVmean, the GCSF dose will be 780 mcg x 1 day
  Interventions: Drug: GCSF
- Phase II-G-CSF (Experimental): Phase 2 participants will be treated with the optimal dose of GCSF found in the phase 1 portion of the study.
  Interventions: Drug: GCSF

INTERVENTIONS:
Drug: GCSF — Granulocyte Colony Stimulating Factor (GCSF)
  Other Names: Filgrastim; Neupogen; Zarxio; G-CSF

SUMMARY:
This is a research study using Granulocyte Colony Stimulating Factor (GCSF) as a bone marrow stimulating agent for imaging to guide radiation treatment planning. G-CSF is a type of growth factor. Growth factors are proteins made in the body. G-CSF is a type of growth factor that makes the bone marrow produce white blood cells to reduce the risk of infection after some types of cancer treatment. GCSF is being given to stimulate the bone marrow to identify the active (blood cell producing regions) to better spare during pelvic radiation treatment planning.

DETAILED DESCRIPTION:
This is a phase 1/2 study. The phase 1 is a dose finding portion of the study and phase 2 will enroll additional patients at the dose found in phase I. Patients in phase I and phase 2 will have the same treatment and follow-up.

Participants will undergo standard of care diagnostic imaging, complete blood count (CBC) with differential and chemistry labs initially. While receiving the GCSF, participants will have a CBC with differential checked a day after each dose and one day prior to first day of radiation. The treatment planning FDG PET/CT will be performed shortly after the GCSF. During chemoradiation, participants will have weekly CBC with differential checked and other labs as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic cancer patients receiving pelvic radiation and chemotherapy, specifically: 1) Stage I-IIIC1 cervix cancer, 2) stage I-III primary vaginal cancer, 3) stage IIIA-IIIC1 endometrial cancer patients status post hysterectomy and lymph node assessment, and 4) recurrent endometrial cancer patients with pelvic confined disease No required para-aortic or extended field radiation
* Age > 18 years
* ECOG performance status 0-2
* Adequate kidney function (serum Cr <1.5 or creatinine clearance >50 mg/dl)
* Adequate bone marrow function (white blood cells > 3.0 X 10^9/L, platelets >100 x 10^9/L)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Treatment for other cancer in the past 2 years
* Previous pelvic radiation
* Medical condition that prevents receiving chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Kidd, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford Cancer Institute Palo Alto, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I -Dose Finding, Cohort 1: Dosing will occur in cohorts of 3 patients with the start at dose of GCSF will be 780 mcg x 2 days.
  FDG PET/CT: Fluorodeoxyglucose (FDG)-positron emission tomography (PET) and computed tomography (CT)
  GCSF: Granulocyte Colony Stimulating Factor (GCSF)
- Phase I -Dose Finding, Cohort 2: Dosing will occur in cohorts of 3 patients, If 3 out of 3 patients achieve the target SUVmean, the GCSF dose will be 780 mcg x 2 days.
  FDG PET/CT: Fluorodeoxyglucose (FDG)-positron emission tomography (PET) and computed tomography (CT)
  GCSF: Granulocyte Colony Stimulating Factor (GCSF)
- Phase I -Dose Finding, Cohort 3: Dosing will occur in cohorts of 3 patients, If 3 out of 3 patients achieve the target SUVmean, the GCSF dose will be 780 mcg x 1 day
  FDG PET/CT: Fluorodeoxyglucose (FDG)-positron emission tomography (PET) and computed tomography (CT)
  GCSF: Granulocyte Colony Stimulating Factor (GCSF)
- Phase II- Phase II-G-CSF: Phase 2 participants will be treated with the optimal dose of GCSF found in the phase 1 portion of the study.
Period: Overall Study
Arm/Group | Phase I -Dose Finding, Cohort 1 | Phase I -Dose Finding, Cohort 2 | Phase I -Dose Finding, Cohort 3 | Phase II- Phase II-G-CSF
Started | 3 | 3 | 1 | 0
Completed | 3 | 3 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I -Dose Finding, Cohort 1: Dosing will occur in cohorts of 3 patients with the start at dose of GCSF will be 780 mcg x 3 days
  FDG PET/CT: Fluorodeoxyglucose (FDG)-positron emission tomography (PET) and computed tomography (CT)
  GCSF: Granulocyte Colony Stimulating Factor (GCSF)
- Phase I -Dose Finding, Cohort 2: Dosing will occur in cohorts of 3 patients, If 3 out of 3 patients achieve the target SUVmean, the GCSF dose will be 780 mcg x 2 days
  FDG PET/CT: Fluorodeoxyglucose (FDG)-positron emission tomography (PET) and computed tomography (CT)
  GCSF: Granulocyte Colony Stimulating Factor (GCSF)
- Total: Total of all reporting groups
Arm/Group | Phase I -Dose Finding, Cohort 1 | Phase I -Dose Finding, Cohort 2 | Phase I -Dose Finding, Cohort 3 | Total
Number analyzed (Participants) | 3 | 3 | 1 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 1 | 6
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 7
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Recommended Phase 2 Dose (RP2D) Criteria
Description: RP2D will be defined as the dose at which the standard uptake value (SUV) on D5 FDG PET reaches a target SUVmean of 2.5 or higher, with normalization of white blood cells (WBC) and absolute neutrophil count (ANC) prior to the start of radiation. The outcome will be reported as the number of participants who meet these criteria.
Time Frame: Up to 1 day after completing GCSF
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I -Dose Finding, Cohort 1 | Phase I -Dose Finding, Cohort 2 | Phase I -Dose Finding, Cohort 3
Number analyzed (Participants) | 3 | 3 | 1
Participants | 3 | 3 | 0

2. Primary Outcome: Number of Participants Experiencing Grade 3 or Greater Neutropenia (ANC < 1000/mm³)
Description: Rate of grade 3 or greater neutropenia (ANC < 1000/mm³ at any point of therapy) was monitored using regular complete blood count (CBC) with differential.
Time Frame: Up to 7 weeks after starting treatment
Measure: Count of Participants; unit: Participants
Groups:
- Phase I - Cohorts 1; Phase I- Cohort 2; Phase I- Cohort 3: GCSF stimulated PET for bone marrow sparring.
  GCSF: Granulocyte Colony Stimulating Factor (GCSF)
Arm/Group | Phase I - Cohorts 1 | Phase I- Cohort 2 | Phase I- Cohort 3
Number analyzed (Participants) | 3 | 3 | 1
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks after treatment.
Arm/Group | Phase I -Dose Finding, Cohort 1 | Phase I -Dose Finding, Cohort 2 | Phase I -Dose Finding, Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I -Dose Finding, Cohort 1 (N=3) | Phase I -Dose Finding, Cohort 2 (N=3) | Phase I -Dose Finding, Cohort 3 (N=1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal Hemmorhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I -Dose Finding, Cohort 1 (N=3) | Phase I -Dose Finding, Cohort 2 (N=3) | Phase I -Dose Finding, Cohort 3 (N=1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)
Pain - Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 3 (7) | 3 (7) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 3 (6) | 2 (7) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (2) | 2 (5) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 3 (5) | 3 (7) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT04514692/Prot_SAP_000.pdf